CLINICAL TRIAL: NCT00836888
Title: ONO-4538 Phase I Study - A Single Center, Open Label, Dose Escalation Single Dose, Followed by Multiple Dose Study of ONO-4538, a Fully Human mAb to PD-1, in Patients With Advanced Malignant Solid Tumors
Brief Title: ONO-4538 Phase I Study in Patients With Advanced Malignant Solid Tumors in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-01
Record Dates: First submitted 2009-01-26; First posted 2009-02-04 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2015-04

CONDITIONS: Malignant Solid Tumor
Keywords: ONO-4538; MDX-1106; solid tumors
MeSH Terms: interventions — Nivolumab

ARMS (1):
- Cohort (Experimental)
  Interventions: Biological: ONO-4538

INTERVENTIONS:
Biological: ONO-4538 — 1mg/kg, 3mg/kg, 10mg/kg and 20mg/kg ONO-4538 infusion cohorts

SUMMARY:
Evaluation of the safety, tolerability and pharmacokinetics (PK) of a single dose and multiple doses of ONO-4538 in Japanese patients with advanced malignant solid tumors, and exploratory evaluation of the pharmacological effect and efficacy of ONO-4538.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of solid tumor with at least one measurable lesion of ≥ 10mm.
* Tumor must be advanced or recurrent which is refractory to standard therapies or for which no alternative, appropriate therapy exists.
* ECOG Performance Status of 0-1
* Life expectancy ≥ 3 months
* Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

* History of severe hypersensitivity reactions to other antibodies.
* Residual adverse reactions or effect of prior therapy, which deemed to affect the safety evaluation of the study drug by the investigator or subinvestigator.
* Two or more synchronous tumors, except for adequately treated basal cell cancer or cancer in situ, or superficial bladder cancer, or any other cancers from which the patient has been disease-free for at least 5 years.
* Patients with any active autoimmune disease or a documented history of chronic or recurrent autoimmune disease, or current medical condition that requires systemic immunosuppressive doses of steroids or other immunosuppressive medications.
* Other exclusion criteria as specified in the study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ohyama Yukiya, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Kanto Region, Kanto, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- ONO-4538 1mg/kg Cohorts: Administer ONO-4538 1mg/kg as an intravenous infusion over ≥1 hour
- ONO-4538 3mg/kg Cohorts: Administer ONO-4538 3mg/kg as an intravenous infusion over ≥1 hour
- ONO-4538 10mg/kg Cohorts: Administer ONO-4538 10mg/kg as an intravenous infusion over ≥1 hour
- ONO-4538 20mg/kg Cohorts: Administer ONO-4538 20mg/kg as an intravenous infusion over ≥1 hour
Period: Overall Study
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Started | 3 | 5 | 6 | 3
Completed | 0 | 2 | 0 | 0
Not Completed | 3 | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts | Total
Number analyzed (Participants) | 3 | 5 | 6 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5 | 1 | 11
  >=65 years | 2 | 1 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 0 | 1 | 7
  Male | 2 | 0 | 6 | 2 | 10
Performance Status（ECOG） [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS 0：Fully active, able to carry on all pre-disease performance without restriction
  1：Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 1 | 1 | 2 | 0 | 4
    1 | 2 | 4 | 4 | 3 | 13
disease stage classification [Count of Participants; unit: Participants] — The stage IV：The cancer has spread to nearby lymph nodes or to organs. The stage IVb：The cancer has spread to distant organs.
  Participants
    IV | 0 | 3 | 0 | 1 | 4
    IVb | 0 | 0 | 2 | 0 | 2
    Recurrent | 3 | 2 | 4 | 2 | 11
Cancer treatment history (surgery) [Count of Participants; unit: Participants]
  None | 0 | 1 | 2 | 2 | 5
  Present | 3 | 4 | 4 | 1 | 12
Cancer treatment history (radiotherapy) [Count of Participants; unit: Participants]
  None | 3 | 3 | 4 | 2 | 12
  Present | 0 | 2 | 2 | 1 | 5
Cancer treatment history (drug therapy) [Count of Participants; unit: Participants]
  None | 0 | 0 | 1 | 0 | 1
  Present | 3 | 5 | 5 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax at Single Dose
Time Frame: day1(before administration, 1 hour after the start of administration, and 2 and 8 hours after the end of administration), day2(24 h), day3(48 h), day4(72 h), day8, day15, and day22 or at the discontinuation
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Number analyzed (Participants) | 3 | 5 | 6 | 3
μg/mL | 24.4 (4.5) | 68.8 (10.9) | 192 (36) | 214 (68)

2. Primary Outcome: AUClast at Single Dose
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg·h/mL
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Number analyzed (Participants) | 3 | 5 | 6 | 3
μg·h/mL | 4950 (580) | 12300 (4500) | 43900 (7200) | 67400 (15500)

3. Primary Outcome: T1/2 at Single Dose
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: day
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Number analyzed (Participants) | 3 | 5 | 6 | 3
day | 15 (0) | 13 (7) | 21 (11) | 17 (9)

4. Primary Outcome: Ceoi at Multiple Doses
Description: Ceoi：Serum concentrations immediately after the end of continuous administration
Time Frame: day 15
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Number analyzed (Participants) | 3 | 5 | 6 | 3
μg/mL | 29.3 (6.0) | 101 (12) | 270 (42) | 286 (112)

5. Secondary Outcome: Best Overall Response
Description: Response Evaluation Criteria In Solid Tumors Criteria (ver 1.0) was used for this Outcome Measure.
  Please see the reference for the detailed description. Therasse, Arbuck et al. New guidelines to evaluate the response to treatment in solid tumors. J Natl Cancer Inst 2000;92:205-16.
Time Frame: up to study completion, every 4 weeks in principle
Measure: Count of Participants; unit: Participants
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
Number analyzed (Participants) | 3 | 5 | 6 | 3
Participants
  CR | 0 | 1 | 0 | 0
  PR | 1 | 0 | 1 | 0
  SD | 0 | 1 | 2 | 0
  PD | 2 | 3 | 3 | 3
  Unknown | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All subjects treated with the study drug were followed up for at least 28 days after the last dose.
Arm/Group | ONO-4538 1mg/kg Cohorts | ONO-4538 3mg/kg Cohorts | ONO-4538 10mg/kg Cohorts | ONO-4538 20mg/kg Cohorts
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5 | 2/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 1mg/kg Cohorts (N=3) | ONO-4538 3mg/kg Cohorts (N=5) | ONO-4538 10mg/kg Cohorts (N=6) | ONO-4538 20mg/kg Cohorts (N=3)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4538 1mg/kg Cohorts (N=3) | ONO-4538 3mg/kg Cohorts (N=5) | ONO-4538 10mg/kg Cohorts (N=6) | ONO-4538 20mg/kg Cohorts (N=3)
Atrial fiblillation (Cardiac disorders) | 0 | 0 | 1 | 0
Venticular extrasystoles (Cardiac disorders) | 0 | 1 | 2 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 2 | 1
Malaise (General disorders) | 0 | 0 | 2 | 1
Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Ammonia increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 1 | 3 | 2 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 3 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 1
Blood uric acid increrased (Investigations) | 0 | 1 | 3 | 1
C-reactive protein increased (Investigations) | 1 | 2 | 2 | 2
Eosinophil count increased (Investigations) | 2 | 3 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 1
Haematocrit decreased (Investigations) | 1 | 3 | 2 | 0
Haematocrit increased (Investigations) | 0 | 0 | 1 | 0
Blood urine preasent (Investigations) | 1 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 3 | 2 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 5 | 2
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 3 | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 3 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 1 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 1 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 1 | 1
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 1
Rheumatoid factor increased (Investigations) | 0 | 1 | 1 | 0
Blood alkaline phosphatese increased (Investigations) | 0 | 1 | 1 | 1
Interleukin level increased (Investigations) | 1 | 0 | 0 | 0
Antinuclear antibody increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypoaeshesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Phrenic nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dematitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Palmar-plantar erythodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes